CLINICAL TRIAL: NCT01582490
Title: Evaluation of the Safety and Efficacy of EXPAREL® (Bupivacaine Liposome Injectable Suspension) When Administered Via Infiltration Versus Instillation in Subjects Undergoing Bilateral Augmentation Mammoplasty
Brief Title: Study of EXPAREL in Patients Undergoing Breast Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA402S23B901
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-05

CONDITIONS: Mammoplasty; Postoperative Pain
Keywords: Mammoplasty; Postoperative pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infiltration - EXPAREL (Active Comparator): Group 2 will receive diluted EXPAREL (i.e., the contents of one 20 mL vial, 266 mg, diluted with 20 mL of preservative-free 0.9% normal saline to a total of 40 mL) for postsurgical analgesia. Half of the resulting mixture (i.e., 20 mL) will be administered via local infiltration into each surgical site per the surgeon's normal practice at the beginning of surgery.
  Interventions: Drug: Instillation - EXPAREL
- Instillation - EXPAREL (Experimental): Group 1 will receive diluted EXPAREL (i.e., the contents of one 20 mL vial, 266 mg, diluted with 20 mL of preservative-free 0.9% normal saline to a total of 40 mL) for postsurgical analgesia. Half of the resulting mixture (i.e., 20 mL) will be instilled into each breast pocket at the beginning of surgery.
  Interventions: Drug: Infiltration - EXPAREL

INTERVENTIONS:
Drug: Instillation - EXPAREL — Intravenous (IV) morphine sulfate, hydromorphone, or oral oxycodone with acetaminophen (5/325 mg) will be permitted following surgery, as needed.
  Other Names: bupivacaine liposomal injectable suspension
  Arms: Infiltration - EXPAREL
Drug: Infiltration - EXPAREL — IV morphine sulfate, hydromorphone, or oral oxycodone with acetaminophen (5/325 mg) will be permitted following surgery, as needed.
  Other Names: bupivacaine liposomal injectable suspension
  Arms: Instillation - EXPAREL

SUMMARY:
This is a Phase 4, prospective, open-label, non-randomized, sequential study with two treatment groups differing only in the technique used for EXPAREL administration (instillation or infiltration).

DETAILED DESCRIPTION:
Each subject underwent bilateral augmentation mammoplasty and received the same dose of EXPAREL. This primary objective of this study was to assess the efficacy of EXPAREL when administered via infiltration versus instillation as part of bilateral augmentation mammoplasty. The secondary objectives were to further assess other efficacy measures and the safety profile of EXPAREL.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-75 years of age inclusive.
* American Society of Anesthesiologists (ASA) physical status 1-3.
* Undergoing bilateral augmentation mammoplasty without any concurrent surgical procedure(s).
* Physically and mentally able to participate in the study and complete all study assessments.
* Able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the study components.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics.
* Any subject whose anatomy or surgical procedure might, in the opinion of the Investigator, preclude the potential successful local administration of EXPAREL.
* Subjects currently pregnant or who may become pregnant during the course of the study.
* Any subject who in the opinion of the Investigator might be harmed or be a poor candidate for participation in the study.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Del Vecchio, MD, Principal Investigator — Steward Research
Locations (1):
- Steward St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Infiltration - EXPAREL: Subjects received EXPAREL 266 mg via infiltration.
- Instillation - EXPAREL: Subjects received EXPAREL 266 mg via instillation.
Period: Overall Study
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Started | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 19 subjects were enrolled, 9 in the Infiltration - EXPAREL group and 10 in the Instillation - EXPAREL group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (7.25) | 29.7 (11.41) | 28.8 (9.57)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
ASA Classification [Number; unit: participants] — There were 19 subjects enrolled. 8 subjects in the Infiltration - EXPAREL group were in the safety analysis set. 10 subjects in the Instillation - EXPAREL group were in the safety analysis set. ASA Class 1 is defined as a normal healthy subject; ASA Class 2 is defined as a subject with mild systemic disease.
  participants
    ASA Class 1 | 5 | 9 | 14
    ASA Class 2 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Description: The primary outcome measure is the duration of analgesia, measured by the time (hours) from the end surgery to the subject's first postsurgical opioid administration.
Time Frame: 10 days
Population: Of the 8 subjects in the Infiltration - EXPAREL group (efficacy analysis set), 5 were censored, leaving 3 subjects who were administered an opioid. Of the 9 subjects in the Instillation - EXPAREL group (efficacy analysis set), 7 were censored, leaving 2 subjects who were administered an opioid.
Measure: Number; unit: hours
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 3 | 2
hours
  Minimum time to postsurgical opioid | 0.07 | 0.3
  Maximum time to postsurgical opioid | 4.28 | 4.82

2. Secondary Outcome: Total Postsurgical Opioid Consumption in the Surgical Center
Description: Total amount of opioids (morphine-equivalent mg) administered postsurgically in each group.
Time Frame: 10 days
Population: There were 8 subjects in the Infiltration - EXPAREL efficacy analysis set and 9 subjects in the Instillation - EXPAREL efficacy analysis set.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
mg | 4.5 (6.26) | 3.0 (7.74)

3. Secondary Outcome: Pain Intensity Assessment Upon Waking in the PACU
Description: Subject-reported pain assessment upon waking in the PACU on a scale of 0 to 10 where 0 = no pain and 10 = worst possible pain.
Time Frame: Upon waking in the PACO post surgery
Population: There were 9 subjects in the Infiltration - EXPAREL efficacy analysis set and 8 subjects in the Instillation - EXPAREL efficacy analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Infiltration - EXPAREL: Subjects received 266 mg EXPAREL via infiltration
- Instillation - EXPAREL: Subjects received 266 mg EXPAREL via instillation
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
units on a scale | 4.5 (2.98) | 3.7 (2.6)

4. Secondary Outcome: Pain Intensity Assessment at the Time of Hospital Discharge
Description: Subject-reported pain assessment at the time of hospital discharge (assessed an average of 3.11 hours after surgery for the Instillation group and 3.20 hours after surgery for the Infiltration group) on a scale from 0 to 10 where 0 = no pain and 10 = worst possible pain.
Time Frame: At the time of hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
units on a scale | 3.8 (1.39) | 3.4 (1.88)

5. Secondary Outcome: Time to Hospital Discharge Being Written
Description: The time (hours) to the hospital discharge being written for subjects in each group,
Time Frame: At the time of hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
hours | 3.2 (0.941) | 3.11 (1.005)

6. Secondary Outcome: Incidence of Opioid-Related Adverse Events
Description: The incidence of adverse events that were assessed as opioid-related
Time Frame: Through 10 Days Post Surgery
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
participants | 0 | 0

7. Secondary Outcome: Overall Rating of Subject Satisfaction With Postsurgical Pain Control at Hospital Discharge
Description: Subject-reported satisfaction with postsurgical pain control in the categories of "extremely dissatisfied," "dissatisfied," "neither satisfied nor dissatisfied," "satisfied," and "extremely satisfied."
Time Frame: At the time of hospital discharge
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
participants
  Extremely Dissatisfied | 1 | 0
  Dissatisfied | 1 | 0
  Neither Satisfied nor Dissatisfied | 0 | 2
  Satisfied | 3 | 3
  Extremely Satisfied | 3 | 4

8. Secondary Outcome: Overall Rating of Subject Satisfaction With Postsurgical Pain Control at Day 10
Description: as for outcome 7
Time Frame: Day 10 after surgery
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Number analyzed (Participants) | 8 | 9
participants
  Extremely Dissatisfied | 2 | 0
  Dissatisfied | 1 | 0
  Neither Satisfied nor Dissatisfied | 1 | 2
  Satisfied | 2 | 2
  Extremely Satisfied | 2 | 5

ADVERSE EVENTS:
Time Frame: From surgery through Day 10.
Arm/Group | Infiltration - EXPAREL | Instillation - EXPAREL
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No